

Chief Investigator: Dr James Stacey, Consultant Clinical Psychologist, Oxfordshire CAMHS Neurodevelopmental Conditions pathway

## Investigating the clinical utility of the Oxford Virtual Autism Assessment Tool (OVAAT)

IRAS Reference: 23/SW/0093

If you would like to take part in the study, please complete the consent form below:

| | Please initial box |
|---|---|
| 1. | I confirm that I have read the information sheet dated 11.09.2023 (Version 2) for the |
| | above study. I have had the opportunity to consider the information, ask questions |
| | and have had these answered satisfactorily. |
| 2. | I understand that I do not have to take part in the study and that it is my choice. I |
| | know that I can stop at any time without telling researchers or staff in the NDC |
| | pathway why. I understand that participating or not participating in the study will not |
| | affect my CAMHS support I may need (now or in future) in any way. |
| 3. | I understand that: |
| | (a) The information I provide as part of this study will be kept confidential and that |
| | the only exception would be if the researchers were concerned that I, or someone |
| | else, might be at risk of serious harm, |
| | (b) If my confidentiality needs to be broken, every effort will be made to discuss this |
| | with me (unless this would e.g., increase the risk of serious harm), |
| | (c) If there is a significant risk of harm to me or someone else, only people who need |
| | to be informed of the risk (i.e., those who can help reduce the risk) will be |
| | informed (e.g. GP, emergency services, CAMHS professionals, parents/caregivers) |
| | and they will only be provided with information relevant to the risk. |
| | (d) I will be informed of what information has been shared, and with whom. |
| 4. | I understand that data collected during the study may be looked at by individuals from |
| | regulatory authorities or from the NHS Trust, where it is relevant to my taking part in |
| | this research. I give permission for these individuals to access data collected about me |
| | during the study. |
| 5. | I understand that I will need to provide a form of identification (e.g. passport, birth certificate, (provisional) driving licence) when I meet a member of the study team for |
| | the OVAAT. |

| 6. | I agree to the OVAAT session being audio and video recorded as part of the research study. | |
|---|---|---|
| 7.<br>8. | I understand that the research team will hold my personal details (e.g., name, contact details) for the duration of the study, in order to contact me for research purposes, and that following completion of the study, this information will be destroyed. I agree to take part in the study. | _ |
| To be | e completed by participant: | |
| Name | e of Participant: | |
| Date: | : | |
| Signa | ature: | |
| <u>NB</u> : Y | ou do not need to provide a signature if you return this form from your or your parent's e-ma | il |
| addre | ess. By returning this form via e-mail (with or without a signature) you will be consenting to tal | ke |
| part i | in the study. | |
| For st | tudy team only: | |
| Name | e of person taking consent: | |
| Date: | : | |
| Signa | ature: | |